CLINICAL TRIAL: NCT05482906
Title: Individual Gait Pattern and MRI Lesion Load to Quantify Gait Impairment in MS: A Cross Sectional Study.
Brief Title: Common and Specific Information From Neuroimaging and Smartphone
Acronym: MS-CSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0203
Record Dates: First submitted 2022-07-20; First posted 2022-08-01 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis
Keywords: Wearable sensor; Gait; MRI
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: eGait — IMU sensor (as part of eGait device) worn at the hip during T25FW
  Other Names: Wearable sensor

SUMMARY:
Gait alteration is frequent in MS and limitation in walking ability is a major concern in MS patients. Umanit and LMJL (Nantes university) has developed a device call egait to assess walking ability in individuals (eg MS patients).

DETAILED DESCRIPTION:
This device consists in a commercialized IMU sensor (MetaMotionR Sensor, Mbientilab) worn at the right hip, a smartphone app and dedicated algorithm/mathematical model to extract raw sensor data and calculate individual gait pattern (IGP). This IGP consists of a curve, based on quaternion and representing the rotation recorded by the IMU during an average gait cycle. Pursue previous works conducted on (IGP to assess) gait alteration in MS by adding (to IGP) new information from MRI.

ELIGIBILITY:
Inclusion Criteria :

* Diagnosis of MS based on McDonald criteria (including Relapsing-remitting and progressive MS)
* Over 18 years old /age greater than 18 years
* Patients followed at Nantes university hospital or Rennes university hospital
* Last known EDSS before inclusion ranging from 0 to 6 inclusive/EDSS of 0 to 6 inclusive, prior inclusion
* No relapse within 3 months
* With a Medullar MRI planed as part as usual care
* Affiliated person or beneficiary of a social security scheme

Exclusion Criteria :

* Bilateral aid needed to walk
* Women who are pregnant
* Patient having expressed their opposition
* Patient under guardianship or security measure

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: MS patients cohort followed at Nantes university hospital or Rennes university hospital (OFSEP HD cohort)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Clustering analyze based on IGP | At the inclusion
  IGP consists of a curve, based on quaternion and representing the rotation recorded by the IMU during an average gait cycle (0-1).
Clustering analyze based on EDSS score | At the inclusion
  EDSS is an ordinal scale measuring disability and ranging from 0 (normal examination) to 10 (death due to MS) in a 0,5-point increments from score 1.
Clustering analyze based on MRI lesion load | At the inclusion
  MRI characteristics are spinal and extraspinal lesion volumes.

SECONDARY OUTCOMES:
Correlation with disability | At the inclusion
  Correlation of IGP obtained during a walk of 25 feet with Expanded Disability Status Scale (EDSS). EDSS is an ordinal scale measuring disability and ranging from 0 (normal examination) to 10 (death due to MS) in a 0,5-point increments from score 1. Here EDSS of 0 to 2 inclusive defined as mild, 2,5 to 4 inclusive as moderate and EFDSS of 4,5 to 6 inclusive defined as severe
Correlation with MRI lesion load | At the inclusion
  Add lesion load (Spinal and extraspinal lesion volume) from MRI to previous correlation.
Building a predictive model for lesion load involving in walk ability from IGP | At the inclusion
  Root mean square error between observed and lesion load predicted by the model, calculated by cross-validation.
Building a predictive model for group belonging from group established in main outcome based on IGP | At the inclusion
  Multiclass accuracy between real and predict group, calculated by cross-validation

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: No